CLINICAL TRIAL: NCT00433680
Title: Targeted Obesity Prevention Program for Adolescent Females
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Research Institute (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DK72932; R01DK072932 (NIH)
Record Dates: First submitted 2007-02-09; First posted 2007-02-12 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-04

CONDITIONS: Obesity
Keywords: adolescent; female; obesity; body dissatisfaction
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Healthy Weight — 4 weekly 1 hour meetings that encourage reductions in fat and sugar intake and increases in physical activity to decrease onset of obesity and body dissatisfaction.
  Other Names: Healthy Weight Project

SUMMARY:
The purpose of this study is to evaluate the effectiveness of an obesity prevention program when administered to female college freshmen.

DETAILED DESCRIPTION:
The goal of this project is to conduct a large randomized controlled trial of a selected obesity prevention program that reduced risk for future onset of obesity over a 2-year follow-up and decreased bulimic symptoms and negative affect in a preliminary trial (N = 188). The Healthy Weight program targets female adolescents with body image concerns because they are a group at high risk for obesity onset. We propose to focus on body-dissatisfied females during the first year of college because this is a particularly high-risk developmental period for weight gain (Butler, Black, Blue, & Gretbeck, 2004; Hovell, Mewborn, Randle, & Fowler-Johnson, 1985). This intervention utilizes persuasion principles from social and clinical psychology (e.g., strategic self-presentation, motivational interviewing) to increase the likelihood that participants will make behavioral changes. This study consists of two components:

We plan to include 405 female college freshmen (aged 17-19) as participants in this study. All first-year female University of Oregon students are mailed a letter of invitation to participate. Posters and flyers on campus are also used as recruitment tools. Participants are assigned to either a healthy weight management condition or a media literacy condition (in which participants learn tricks media use to enhance women's appearance). In both conditions, participants attend four weekly 1-hour sessions led by female research assistants from the Oregon Research Institute. All participants complete 5 structured psychiatric interviews assessing current Diagnostic and Statistical Manual (DSM-IV) symptoms of anorexia nervosa, bulimia nervosa, and binge eating disorder, as well as psychiatric conditions that commonly co-occur with bulimia nervosa during adolescence. Participants also complete 5 surveys that focus on her attitudes, feelings, and behaviors over the past month. Surveys and interviews are administered by trained assessors at baseline, one month later, 6 months from baseline, 12 months from baseline, and 24 months from baseline. Participants' height and weight are also measured during these assessments. If a participant meets criteria for an eating disorder at any assessment point, she is told in a clinically sensitive fashion that a more intensive intervention is needed and treatment referrals are provided. If a participant meets criteria for a co-morbid condition, she is informed of the need to seek treatment, but she is allowed in the study. If a participant is already very thin (in the lowest 5th percentile weight for her height), she is told that it may be dangerous to participate in an intervention that might result in further weight loss, and she will not be allowed in the study. Participants are paid for completing the assessments ($30 for completing each survey and interview, with a $30 bonus for completing all assessments, for a total of $180 over the course of two years). Participants randomly selected to participate in the Validity Sub-study (described below) have the opportunity to earn an additional $180. Identifying information never appears on any interviews or surveys. Identifying information will be collected on separate forms for tracking purposes only. Interviews, surveys, and identifying information forms are transported immediately to Oregon Research Institute by trained assessors.

We will conduct an intensive validation substudy with a randomly selected 15% of participants (n = 60). We plan to assess the validity of self-reported caloric intake with doubly labeled water, and the validity of self-reported activity levels with tri-axial accelerometers. We will also measure resting metabolic rate using a ventilated hood. For each of the 2 academic quarters that we recruit participants during each of the 3 proposed recruitment years, 10 participants will be randomly selected to provide intensive data during the last 2 weeks of the interventions because this should be the period during which there is maximal difference between participants in the two conditions in terms of caloric intake and physical activity. Participants in the validity sub-study will complete all assessments in the University of Oregon's human physiology lab. Assessments will be carried out by trained human physiology staff. Participants will complete pregnancy tests prior to participating in the validity substudy. Pregnant participants will not be able to complete the validity substudy as an extra precaution against any risk to the fetus that may be posed by the doubly labeled water procedure. No risks to fetuses or pregnant women from doubly labeled water have been identified at this point in time. Participants in this substudy will complete a 4-hour assessment within 2 days after the second intervention session (week 2) and will complete another 2-hour assessment within 2 days after the fourth intervention session. Participants will be offered an additional $80 for coming to the lab for the first 4-hour assessment and $100 for coming to the lab for the second 2-hour assessment.

ELIGIBILITY:
Inclusion Criteria:

* All female college freshmen at the University of Oregon will be invited to participate in the study.

Exclusion Criteria:

* Any participant that meets criteria for an eating disorder at any assessment point will be excluded from the study.
* Any participant with BMI below 5% for their age group will be excluded to avoid health risks
* Any participant who does not report some form of body dissatisfaction will be excluded from the study

Ages: 17 Years to 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 405 (Estimated)
Dates: Start 2007-03; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
risk for future onset of obesity and weight gain | 2 years

SECONDARY OUTCOMES:
measure changes in caloric intake, physical activity, and body dissatisfaction | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Eric Stice, PhD, Principal Investigator — Oregon Research Institute
Locations (1):
- Oregon Research Institute, Eugene, Oregon, United States

REFERENCES:
- [Result] Stice E, Sysko R, Roberto CA, Allison S. Are dietary restraint scales valid measures of dietary restriction? Additional objective behavioral and biological data suggest not. Appetite. 2010 Apr;54(2):331-9. doi: 10.1016/j.appet.2009.12.009. Epub 2009 Dec 16. PMID 20006662
- [Derived] Rohde P, Arigo D, Shaw H, Stice E. Relation of self-weighing to future weight gain and onset of disordered eating symptoms. J Consult Clin Psychol. 2018 Aug;86(8):677-687. doi: 10.1037/ccp0000325. PMID 30035584
- [Derived] Stice E, Palmrose CA, Burger KS. Elevated BMI and Male Sex Are Associated with Greater Underreporting of Caloric Intake as Assessed by Doubly Labeled Water. J Nutr. 2015 Oct;145(10):2412-8. doi: 10.3945/jn.115.216366. Epub 2015 Sep 2. PMID 26338886
- [Derived] Stice E, Durant S. Elevated objectively measured but not self-reported energy intake predicts future weight gain in adolescents. Appetite. 2014 Oct;81:84-8. doi: 10.1016/j.appet.2014.06.012. Epub 2014 Jun 12. PMID 24930597
- [Derived] Stice E, Durant S, Burger KS, Schoeller DA. Weight suppression and risk of future increases in body mass: effects of suppressed resting metabolic rate and energy expenditure. Am J Clin Nutr. 2011 Jul;94(1):7-11. doi: 10.3945/ajcn.110.010025. Epub 2011 Apr 27. PMID 21525201